CLINICAL TRIAL: NCT05121168
Title: Continuous Erector Spinae Plane Blocks to Treat Pain Following Percutaneous Nephrolithotomy: A Randomized, Placebo-controlled Clinical Trial
Brief Title: Continuous Erector Spinae Plane Blocks to Treat Pain Following Percutaneous Nephrolithotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCNL and cESPB
Record Dates: First submitted 2021-11-04; First posted 2021-11-16 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Pain, Acute Postoperative; Renal Stone
MeSH Terms: conditions — Pain, Postoperative; Nephrolithiasis

STUDY DESIGN:
Intervention Model Description: Randomized, Triple-Masked, Placebo-Controlled, Parallel-Arm Human Subjects Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All individuals other than the investigational pharmacist who prepares each infusion pump reservoir will be masked to treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active Treatment (Experimental): Administration of bupivacaine 0.25% through a perineural catheter inserted into the erector spinae plane (programmed intermittent bolus of 21 mL every 4 hours and no patient-controlled bolus)
  Interventions: Drug: Active bupivacaine 0.25% via an erector spinae plane perineural catheter
- Placebo (Placebo Comparator): Administration of normal saline through a perineural catheter inserted into the erector spinae plane (programmed intermittent bolus of 21 mL every 4 hours and no patient-controlled bolus)
  Interventions: Drug: Placebo normal saline via an erector spinae plane perineural catheter

INTERVENTIONS:
Drug: Active bupivacaine 0.25% via an erector spinae plane perineural catheter — Administration of bupivacaine 0.25% through a perineural catheter inserted into the erector spinae plane (programmed intermittent bolus of 21 mL every 4 hours and no patient-controlled bolus)
  Arms: Active Treatment
Drug: Placebo normal saline via an erector spinae plane perineural catheter — Administration of normal saline through a perineural catheter inserted into the erector spinae plane (programmed intermittent bolus of 21 mL every 4 hours and no patient-controlled bolus)
  Arms: Placebo

SUMMARY:
This is a randomized, triple-masked, placebo-controlled parallel-arm human subjects clinical trial investigating the addition of a continuous erector spinae plane nerve block to a single-injection erector spinae plane block to provide postoperative analgesia following percutaneous nephrolithotomy. Participants will all receive a single-injection nerve block and perineural catheter insertion. Following surgery, participants will be randomly allocated to receive either perineural local anesthetic or normal saline until the second day following surgery.

DETAILED DESCRIPTION:
Enrollment. Participants will be consenting adults undergoing percutaneous nephrolithotomy. Study inclusion will be proposed to eligible patients prior to surgery. If a patient desires study participation, written, informed consent will be obtained. The study population of interest includes women and men of all races, ethnicity, sexual identity, and socioeconomic status. Of note, the investigators will be using local anesthetic, perineural catheters, and infusion pumps as approved/cleared and do not plan to research a possible change of indication or use of these medications/devices as part of this research project.

Preoperative Procedures. Following written, informed consent, the investigators will record baseline anthropometric information (age, sex, height, weight, stone size/burden, comorbidities, prior stone history, glomerular filtration rate, and current stone location and burden) that is already provided by all patients having surgery. Participants will have a peripheral intravenous (IV) catheter inserted, standard noninvasive monitors applied, supplemental oxygen administered via a nasal cannula or face mask and positioned sitting. Midazolam and fentanyl (IV) will be titrated for patient comfort, while ensuring that patients remain responsive to verbal cues. The area of insertion on the ipsilateral side as the surgery will be sterilely prepared, and a clear, sterile, fenestrated drape applied. With ultrasound guidance after subcutaneous local infiltration with lidocaine, a 17g Tuohy and 5-10 ml of saline with 1:200,000 epinephrine will be used to identify the correct plane, as defined by a hyperechoic shadow of the 8th transverse process and erector spine muscle immediately superficial. Once appropriate needle tip location is confirmed, a perineural catheter will be inserted under ultrasound guidance.

Following negative aspiration, 20 mL of 0.25% bupivacaine with 1:200,000 of epinephrine will be injected via the catheter with sonographic confirmation of local anesthetic spread. Blocks will be considered successful if, within 30 minutes, the participant experiences decreased sensation to cold temperature over the level of the ipsilateral 8th thoracic dermatome at the level of anterior axillary line. Failed blocks/catheters will be successfully replaced, or the participant withdrawn from the study.

Treatment Group Assignment. Each participant will be randomized to one of two treatment groups: bupivacaine 0.25% or normal saline ("study infusate").

Randomization will be stratified by surgeon, in block sizes of 4. The randomization list will be created by the University of California San Diego Investigational Drug Service. Investigational pharmacists will prepare all study solutions as determined by the randomization list. Bupivacaine and normal saline are indistinguishable in appearance, and therefore investigators, participants, and all clinical staff will be masked to treatment group assignment for the duration of the enrollment and data collection period. Unmasking will not occur until statistical analysis is complete (termed "triple masking").

Study intervention. Perineural study infusate administration will be initiated within the operating or recovery rooms. The infusion pump will be programmed to deliver an automatic intermittent bolus of 21 mL every 4 hours and no patient-controlled bolus (300 mL reservoir). This dose of bupivacaine is well-within the standard maximum dose at the University of California San Diego for perineural local anesthetic administration for other truncal locations such as the paravertebral space. For any cases of inadvertent premature catheter dislodgement, the subject may opt to have the catheter replaced if logistically possible.

Participants will be discharged home when ready, as determined by standard criteria by the masked surgical service. Perineural catheters will be removed by patient caretakers upon study infusate reservoir exhaustion (approximately 55 hours).

Postoperative analgesics. In addition to the perineural study infusate, subjects will receive standard-of-care oral and intravenous postoperative analgesics which can include acetaminophen, ibuprofen, ketorolac, and opioids (this is surgeon- and patient-dependent). Therefore, all patients of this study-regardless of the treatment arm they are randomized to-will continue to receive current usual and customary analgesia: all will receive the same combination of acetaminophen, ibuprofen, ketorolac, opioids, and a single-injection erector spinae plane block as they would regardless of study participation.

Statistical Methods. The overall objective of the proposed research is to determine the risks and benefits of adding a continuous erector spinae plane (ESP) block to a single-injection ESP in patients undergoing percutaneous nephrolithotomy.

Specific Aim: To determine the benefits and risks of adding a continuous ESP block to the current standard-of-care treatment of a single-injection ESP block and oral opioids following percutaneous nephrolithotomy.

Compared with a single-injection ESP block following percutaneous nephrolithotomy…

Hypothesis 1 [primary]: The addition of a multiple-day continuous ESP block will decrease the severity of pain over the two days following surgery (as measured on the 11-point numeric rating scale).

Hypothesis 2 [primary]: The addition of a multiple-day continuous ESP block will decrease cumulative opioid consumption over the two days following surgery (as measured in oral oxycodone equivalents).

Primary outcome: To claim that the addition of an ambulatory continuous ESP block is superior to a single-injection ESP block alone, at least one of the first 2 hypotheses must be superior while the other at least non-inferior.

Hypothesis 3: The addition of a multiple-day continuous ESP block will decrease the maximum daily severity of pain during the two days following surgery (as measured on the 11-point numeric rating scale).

Hypothesis 4: The addition of a multiple-day continuous ESP block will decrease the number of sleep disturbances due to pain during the second night following surgery.

Hypothesis 5: The addition of a multiple-day continuous ESP block will decrease pain's interference with physical and emotional functioning the day following surgery (as measured with the Interference subscale of the Brief Pain Inventory, Short Form).

Analysis Approach Baseline characteristics by randomized group (bupivacaine vs placebo) will be summarized with means, standard deviations, and quartiles. Balance between groups will be assessed. Specifically, standardized differences will be calculated using Cohen's d whereby the difference in means or proportions is divided by the pooled standard deviation estimates. Any key variables (age, sex, height, weight, and body mass index) with an absolute standardized difference >0.78 (with 1.96×√(2/25)=0.554 [with a sample size of 50, we expect about 25 randomized to bupivacaine vs placebo]) will be noted and included in a linear regression model to obtain an estimate of the treatment effect adjusted for the imbalanced covariate(s). If residuals from the linear regression indicate violations of key assumptions (i.e. homoscedasticity or Gaussian distribution), data transformations and/or alternative generalized linear models will be applied as appropriate. If no imbalance is detected, the primary analysis will proceed by a two-sample Mann-Whitney test. Secondary outcomes will also be analyzed by Mann-Whitney test, or linear models (or generalized linear models) as appropriate to adjust for any imbalanced covariates.

Gatekeeping strategy Again, to claim that the addition of an ambulatory continuous ESP block is superior to a single-injection ESP block alone, at least one of the first 2 hypotheses must be superior while the other at least non-inferior. Additional hypotheses will be tested with strong control of the family-wise error rate at 5%. Testing begins with co-primary hypotheses H1 and H2. If a given test does not reach local significance, alpha is spent and cannot be passed along to hypotheses further along the graph. Otherwise, alpha is not spent and is passed along.

Simulated Power for Numeric Rating Scale for Pain Power is estimated by the following: Numeric Rating Scale difference scores are distributed with a median (interquartile range) of 3 (2 to 4) for placebo and 2 (1 to 3) for active. A sample size of n=25 individuals per group will provide 82% power to detect such an effect with two-sided α=0.05.

Simulated Power for cumulative opioid consumption over the two days Similarly assuming the standard deviation of opioid consumption is about 1 mg, a sample size of n=25 individuals per group will provide 92% power to detect a group difference of 1 mg with two-sided α=0.05.

ELIGIBILITY:
Inclusion Criteria:

* undergoing unilateral percutaneous nephrolithotomy in the prone position
* analgesic plan includes a single-injection erector spinae plane block
* age 18 years or older

Exclusion Criteria:

* morbid obesity as defined by a body mass index > 40 (BMI=weight in kg / [height in meters]2)
* renal insufficiency (abnormal preoperative creatinine or estimated glomerular filtration rate)
* chronic opioid use (daily use within the 2 weeks prior to surgery and duration of use > 4 weeks)
* history of opioid abuse
* any comorbidity which results in moderate or severe functional limitation
* inability to communicate with the investigators or hospital staff
* pregnancy
* bilateral or multi-stage surgical procedures
* incarceration
* known allergy to any study medication
* any contraindication to perineural catheter insertion (e.g., infection at the catheter insertion site)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2025-11-06 (Actual); Study Completion 2025-11-08 (Actual)

PRIMARY OUTCOMES:
The mean of the "average" pain at rest on postoperative days 1 and 2 as measured using the numeric rating scale, collected on postoperative days 1 and 2 | From discharge from the recovery room until the data collection phone call on postoperative day 1, and for the previous 24 hours of the data collection phone call on postoperative day 2.
  The numeric rating scale is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale. To claim that the addition of an ambulatory continuous erector spinae plane block is superior to a single-injection block alone, at least one of the two primary outcomes must be superior while the other at least non-inferior.
Total opioid consumption from recovery room discharge until the data collection phone call on postoperative day 2 (measured in oral oxycodone equivalents) | From recovery room discharge until the data collection phone call on postoperative day 2
  Total opioid consumption from recovery room discharge until the data collection phone call on postoperative day 2 (measured in oral oxycodone equivalents). To claim that the addition of an ambulatory continuous erector spinae plane block is superior to a single-injection block alone, at least one of the two primary outcomes must be superior while the other at least non-inferior.

SECONDARY OUTCOMES:
"Worst" pain as measured using the numeric rating scale | 3 time points queried on postoperative days 1-3: from recovery room discharge through the data collection phone call on postoperative day 1; and then the 24 hours preceding a data collection phone call on each of postoperative days 2 and 3
  The numeric pain scale is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale
"Worst" pain specifically during urination as measured using the numeric rating scale | 3 time points queried on postoperative days 1-3: from recovery room discharge through the data collection phone call on postoperative day 1; and then the 24 hours preceding a data collection phone call on each of postoperative days 2 and 3
  The numeric pain scale is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale
"Average" pain as measured using the numeric rating scale | 3 time points queried on postoperative days 1-3: from recovery room discharge through the data collection phone call on postoperative day 1; and then the 24 hours preceding a data collection phone call on each of postoperative days 2 and 3
  The numeric pain scale is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale
"Least" pain as measured using the numeric rating scale | 3 time points queried on postoperative days 1-3: from recovery room discharge through the data collection phone call on postoperative day 1; and then the 24 hours preceding a data collection phone call on each of postoperative days 2 and 3
  The numeric pain scale is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale
"Current" pain at the time of the data collection phone call as measured using the numeric rating scale | 3 time points queried on postoperative days 1-3
  The numeric pain scale is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale
Sleep disturbances due to pain | 3 time points queried on postoperative days 1-3
  The number of instances the patient awoke due to pain the previous evening
Opioid consumption | 3 time points queried on postoperative days 1-3: from recovery room discharge through the data collection phone call on postoperative day 1; and then the 24 hours preceding a data collection phone call on each of postoperative days 2 and 3
  Opioid consumption measured in oral oxycodone equivalents
Time until first opioid consumption | Queried at each data collection phone call on postoperative days 1-3
  Time measured in hours from surgical stop until the first use of an opioid analgesic
Brief pain Inventory, short form (interference subscale) | 3 time points queried on postoperative days 1-3: from recovery room discharge through the data collection phone call on postoperative day 1; and then the 24 hours preceding a data collection phone call on each of postoperative days 2 and 3
  The Brief pain Inventory (short form) is an instrument specifically designed to assess pain and its impact on physical and emotional functioning. The brief Inventory is comprised of three domains: (1) pain, with four questions involving "worst", "average" and "current" pain levels using a 0-10 numeric rating scale;(2) percentage of relief provided by pain treatments with one question [reported score is the percentage divided by 10 and then subtracted from 10: 0=complete relief,10=no relief] and, (3) interference with 7 questions involving physical and emotional functioning using a 0-10 Likert scale [0=no interference;10=complete interference]: general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life. This outcome will include the interference subscale.
Hospitalization duration | 3 time points queried on postoperative days 1-3: from recovery room discharge through the data collection phone call on postoperative day 1; and then the 24 hours preceding a data collection phone call on each of postoperative days 2 and 3
  The duration of time from surgical stop until discharge measured in hours
Incidence of returns to the emergency department for pain | From hospital discharge through the data collection call on postoperative day 3
  The percentage of participants in each treatment group who in the first three days return to the emergency department due to pain
Incidence of readmissions due to pain | From hospital discharge through the data collection call on postoperative day 3
  The percentage of participants in each treatment group who in the first three days are readmitted due to pain
Inadvertent catheter dislodgement | From the recovery room through the data collection phone call on postoperative day 3
  The percentage of participants in each treatment group who in the first three days have an inadvertent catheter dislodgement
Surgical start as recorded using military time format | Intraoperative (Within the operating room)
  The time of the surgical incision as recorded using military time format
Surgical stop as recorded using military time format | Intraoperative (Within the operating room)
  The time of the final suture insertion as recorded using military time format
Surgical duration | Intraoperative (Within the operating room)
  The time from surgical start to surgical stop measured in minutes and hours
Wisconsin Stone Quality of Life Questionnaire (WISQOL) scores at baseline and postoperative day 2 | Measured at baseline and postoperative day 2
  The Wisconsin Stone Quality of Life questionnaire (WISQOL) is a disease-specific health-related quality of life (HRQOL) instrument designed to assess the impact on patients of stones in the urinary tract (urolithiasis).
Renal access location | intraoperative
  Anatomic approach to the kidney to establish the percutaneous tract for percutaneous nephrolithotomy with 5 possibilities: lower, mid or upper pole, supracostal vs infracostal

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, MD, MS, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - UC San Diego, San Diego, California
  - University of California, San Diego, San Diego, California

IPD SHARING:
Plan to Share IPD: No